CLINICAL TRIAL: NCT05271279
Title: A Single-Arm, Open-Label, Investigator-Initiated Clinical Trial to Evaluate the Safety, Tolerability and Efficacy of Oncolytic Virus Injection (OVV-01) in Combination With IBR900 Cell Injection in Patients With Advanced Malignant Tumors
Brief Title: A Study of OVV-01 Injection in Combination With IBR900 Cell Injection in Patients With Advanced Malignant Tumors
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Research and development strategy adjustment
Sponsor: Beijing Boren Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BR20210414003
Record Dates: First submitted 2022-02-23; First posted 2022-03-09 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-03

CONDITIONS: Advanced Solid Tumor; Relapsed/Refractory Lymphoma
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OVV-01 Injection+IBR900 Cell Injection (Experimental): OVV-01 injection combined with IBR900 cell injection, 2 dose gradients are used for the OVV-01 injection, and the total infusion dose of IBR900 cell injection is 4.0×10^9 cells per cycle.
  Interventions: Biological: OVV-01 Injection+IBR900 Cell Injection

INTERVENTIONS:
Biological: OVV-01 Injection+IBR900 Cell Injection — 2 dose gradients are used for the OVV-01 injection, and the total infusion dose of IBR900 cell injection is 4.0×10^9 cells per cycle.
  OVV-01 injection will be first administered at W1D1 and then at W4D1 followed by every 2 weeks as a treatment cycle, for a total of 6 doses; after the test in the high-dose group is completed, the investigator and sponsor will determine whether to adjust the dosing frequency of OVV-01 (such as once a week) based on the result evaluations. The IBR900 cell injection will be first administered at W1D3 and W1D5 for 2 infusions, and then at W4D3 and W4D5, followed by every 4 weeks as a cycle, for a total of 4 doses, and cell infusions will be conducted at W1, W4, W8 and W12, respectively.

SUMMARY:
This is a prospective, multi-center, open-label, single-arm, investigator-initiated clinical trial to evaluate the safety and efficacy of oncolytic virus injection (OVV-01) in combination with trained immunity NK (tiNK) cell injection (IBR900) for patients with advanced malignant tumors.

DETAILED DESCRIPTION:
In this study, it is planned to enroll about 6-12 subjects with advanced solid tumors or relapsed/refractory lymphomas who have failed in the third-line or higher standard of care in about 1-3 study sites in China. A 2-dose gradient joint exploratory study using the traditional "3+3" mode is adopted in this study. If the high-dose group does not yet reach the MTD, the investigator and funder will decide whether to continue the dose escalation and whether to add a new dose group.

2 dose gradients are used for the OVV-01 injection, and the total infusion dose of IBR900 cell injection is 4.0×10^9 cells per cycle.

OVV-01 injection will be first administered at W1D1 and then at W4D1 followed by every 2 weeks as a treatment cycle, for a total of 6 doses; after the test in the high-dose group is completed, the investigator and sponsor will determine whether to adjust the dosing frequency of OVV-01 (such as once a week) based on the result evaluations. The IBR900 cell injection will be first administered at W1D3 and W1D5 for 2 infusions, and then at W4D3 and W4D5, followed by every 4 weeks as a cycle, for a total of 4 doses, and cell infusions will be conducted at W1, W4, W8 and W12, respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are ≥18 years old and ≤75 years old, male or female;
2. Subjects with advanced malignant tumors with the primary lesions and/or metastatic lesions diagnosed by histopathology/cytological examinations, including but not limited to: melanoma, the head and neck squamous cell carcinoma, cervical carcinoma, osteosarcoma, nasopharyngeal carcinoma, breast carcinoma, lung carcinoma, colorectal carcinoma, liver carcinoma, gastric carcinoma, lymphoma, etc.;
3. Subjects with solid tumors or relapsed/refractory lymphomas who have failed in the third-line or higher standard of care;
4. Subjects with at least one measurable lesion (non-lymph node lesion with longest diameter ≥10 mm, or lymph node lesion with short diameter ≥15 mm) according to the Response Evaluation Criteria in Solid Tumors (RECIST 1.1) or the Evaluation Criteria for Efficacy of Lymphoma Lugano 2014;
5. Subjects with the Eastern Cooperative Oncology Organization (ECOG) score of 0-2;
6. Subjects with the expected survival ≥ 3 months;
7. Subjects with adequate bone marrow function:

   * White blood cell (WBC)≥3.0×10^9/L;
   * Neutrophils (ANC)≥1.5×10^9/L (cannot use the colony stimulating factor within 3 days before the test);
   * Lymphocyte count ≥6.0×10^8/L;
   * Platelet count ≥100×10^9/L;
   * Hemoglobin ≥9.0 g/dL;
8. Subjects with adequate liver function and kidney function:

   * Total bilirubin ≤1.5 times the upper limit of normal (ULN), or total bilirubin ≤3.0×ULN for subjects with liver metastases.
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT)≤2.5×ULN, or AST and ALT≤5×ULN for subjects with liver metastases;
   * Serum creatinine≤1.5×ULN, or creatinine clearance ≥50 ml/min (calculated according to Cockcroft/Gault formula);
9. Coagulation function

   * For subjects not receiving anticoagulation therapy: international normalized ratio (INR)≤1.5×ULN, activated partial thromboplastin time (APTT)≤1.5×ULN
   * For subjects receiving anticoagulation therapy: INR≤ 2-3×ULN, APTT≤ 2-3×ULN Female subjects of childbearing age who is negative in the pregnancy test within 14 days before inclusion. Female subjects of childbearing age and male subjects whose partners are females of childbearing age must agree to use at least one medically approved birth control (such as surgical sterilization, oral contraceptives, intrauterine devices, sexual desire control or barrier contraception in combination with spermicides, etc.);

11.The subjects should voluntarily participate in the study, sign the informed consent forms, have good compliance, and cooperate with the follow-up visits.

Exclusion Criteria:

1. Subjects without measurable lesions;
2. Subjects with symptomatic brain metastases (but subjects who have asymptomatic brain metastases or have been clinically stable for more than 3 months with local treatment can be included in the study);
3. Subjects who have received radiotherapy for the target lesion within 2 months;
4. Subjects with other active malignant tumors that require simultaneous treatment;
5. Subjects who are known to be allergic to the study drug or its active ingredients and excipients;
6. Subjects who have received or been receiving or still need to receive other investigational drug or antiviral treatments within 4 weeks before administration;
7. Subjects who are going to undergo or have received tissue/organ transplantation;
8. Subjects who have active infections or fever >38.5°C of unknown cause during the screening phase and before the first dose;
9. Subjects with active tuberculosis (TB) who are receiving anti-tuberculosis treatment or have received anti-tuberculosis treatment within 1 year before screening;
10. Subjects who are positive in the treponema pallidum serology test;
11. Subjects with the medical history of known human immunodeficiency virus (HIV) positive or known acquired immunodeficiency syndrome (AIDS);
12. Subjects with active hepatitis. Hepatitis B: HBeAg (+), HBcAb (+) in combination with+ HbsAg (+); for HBsAg (+) or HBcAb (+), the detection value of HBV DNA is ≥1000 IU/ml; hepatitis C: hepatitis C virus antibody (HCV Ab) positive and the detection value of HCV RNA is ≥1000 IU/ml; co-infection of hepatitis B and C;
13. Subjects who have received anti-tumor drug therapy such as chemotherapy, radiotherapy, biological therapy, endocrine therapy, and immunotherapy within 4 weeks before the first administration except the following:

    * nitrosourea or mitomycin C within 6 weeks before the first administration of the study drug;
    * oral fluorouracil and small-molecular targeted drugs within 2 weeks before the first administration of the study drug or 5 half-lives of the drug (whichever is longer);
    * traditional Chinese medicine with anti-tumor indications within 2 weeks before the first administration of the study drug;
14. Subjects with cardiovascular disorders meet any of the following:

    * Congestive heart failure with heart function ≥ New York Heart Association (NYHA) III;
    * Severe arrhythmia requiring drug therapy;
    * Acute myocardial infarction, severe or unstable angina, coronary or peripheral artery bypass, and stent within 6 months before the first administration;
    * Left ventricular ejection fraction (LVEF)< 50%;
    * Corrected QTc interval > 450 ms for male and> 470 ms for female, or risk factors for torsade de pointes ventricular tachycardia, such as clinically significant hypokalemia judged by the investigator, family history of long QT syndrome, or familial arrhythmia history (such as pre-excitation syndrome);
    * Uncontrolled hypertension (defined as systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg with treatment with standardized antihypertensive drugs)
15. Subjects with active autoimmune diseases or a history of autoimmune diseases but may be relapsed; but subjects with the following diseases are not excluded and can be further screened:

    * Type 1 diabetes mellitus;
    * Hypothyroidism (if only hormone replacement therapy can be used to control);
    * Controlled celiac disease;
    * Skin diseases that do not require systemic treatment (such as vitiligo, psoriasis, alopecia);
    * Any other diseases that will not relapse without external triggers;
16. Subjects with any diseases who need to use glucocorticoids (prednisone >10 mg/day or equivalent doses of similar drugs) or other immunosuppressive agents for systemic treatment within 14 days before administration of the study drug, but is using or have used any of the following steroids can be included:

    * Adrenaline replacement steroids (prednisone ≤10 mg/day or equivalent dose of similar drugs);
    * Local, ophthalmic, intra-articular, intranasal or inhaled corticosteroids with minimal systemic absorption;
    * Prophylactically short-term (≤7 days) use of corticosteroids (such as allergy to contrast agents) or for the treatment of non-autoimmune diseases (such as delayed hypersensitivity reactions caused by contact allergens);
17. Subjects with psychiatric disorders, alcoholism, heavy smoking, drug use or drug abuse, etc.;
18. Female subjects who are pregnant or breastfeeding, or who are expected to become pregnant during the study (from the screening visit until 180 days after administration) and male subjects who are expected to conceive their partners;
19. Subjects whose adverse reactions of prior anti-tumor treatments have not yet recovered to CTCAE v5.0 Grade 1 (except for the alopecia);
20. Subjects who have serious uncontrollable diseases or other conditions that may affect the treatment of this study and are not suitable to participate in this study as determined by the investigator.

Other conditions not suitable for enrollment at investigators' decision.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-12-24 (Actual); Primary Completion 2022-08-29 (Actual); Study Completion 2022-08-29 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | 7 weeks after initial administration
  To evaluate the safety and tolerability of OVV-01 injection and IBR900 cell injection
Adverse events (AEs) | 24 weeks after initial administration
  The incidence and severity of AEs assessed according to Common Terminology Criteria for Adverse Events (CTCAE) v5.0, and the correlation between AEs and OVV-01 injection combined with IBR900 cell injection

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to 1 year after administration
  To evaluate the effectivity of OVV-01 injection and IBR900 cell injection
Progression-free survival (PFS) | Up to 1 year after administration
  To evaluate the effectivity of OVV-01 injection and IBR900 cell injection
Overall survival (OS) | Up to 1 year after administration
  To evaluate the effectivity of OVV-01 injection and IBR900 cell injection
Disease control rate (DCR) | Up to 1 year after administration
  To evaluate the effectivity of OVV-01 injection and IBR900 cell injection
Duration of overall response (DOR) | Up to 1 year after administration
  To evaluate the effectivity of OVV-01 injection and IBR900 cell injection
Peak plasma concentration of OVV-01 | 14 days after the last administration
  Blood samples will be collected at specified time points to detect the concentration of OVV-01 in peripheral blood and to evaluate the PK parameters
Peak plasma concentration of IBR900 cells | 16 days after initial administration
  Blood samples will be collected at specified time points to detect the concentration of IBR900 cells in peripheral blood and to evaluate the PK parameters
Plasma concentration of anti-VSV-G antibody and neutralizing antibody | 16 weeks after initial administration
  To observe and evaluate the time, titer, and subject rate of antibody development after administration

CONTACTS AND LOCATIONS:
Overall Officials: Kai Hu, MD/PhD, Principal Investigator — Beijing Boren Hospital
Locations (1):
- Beijing Boren Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No